CLINICAL TRIAL: NCT06913790
Title: Evaluation of Central Corneal Thickness in Patients With Vernal Keratoconjunctivitis Using Topical Steroids
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSRSW/Batch-Fall23/808
Record Dates: First submitted 2025-03-29; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Vernal Keratoconjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective observational cohort study aims to assess changes in central corneal thickness (CCT) in vernal keratoconjunctivitis (VKC) patients using topical steroids. Data will be collected from tertiary care hospitals such as Al-Mustafa eye hospital and Jinnah Hospital, Lahore.

DETAILED DESCRIPTION:
A total of 34 participants, including an adjustment for a 10% dropout rate, will be recruited using purposive sampling. The study will last six months. Eligible participants (aged 5-25 years) must have a confirmed VKC diagnosis and be on topical steroids, with exclusions for prior ocular surgery, systemic steroid use, and contact lens wear. Baseline assessments will include demographic data, VKC severity, and CCT measurements via pachymetry and optical coherence tomography. Follow-up evaluations at one and three months will track CCT changes. A paired t-test will compare baseline and follow-up measurements. This study will help understand the impact of topical steroids on CCT in VKC patients.

ELIGIBILITY:
Inclusion Criteria:

* Young adults aged between 5-25 years
* Confirmed diagnosis of VKC
* Currently prescribe topical steroid e.g, dexamethasone, prednisolone
* No prior history of corneal surgery or trauma
* Willing to attend follow-up visits and comply with the treatment protocol.

Exclusion Criteria:

* History of ocular surgery or trauma
* Presence of other corneal pathologies (e.g., Keratoconus)
* Systemic immunosuppressant use or history of systemic steroid use in the past 06 months
* Use of other medications that could influence corneal thickness e.g, antiglaucoma drugs
* Contact lens use within 1 month prior to the study
* Severe dry eye or another ocular surface disease"

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This prospective observational cohort study aims to assess changes in central corneal thickness (CCT) in vernal keratoconjunctivitis (VKC) patients using topical steroids. Data will be collected from tertiary care hospitals such as Al-Mustafa eye hospital and Jinnah Hospital, Lahore
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Slit Lamp Test | 12 Months
  A slit lamp exam, a common eye test, uses a microscope and a focused light beam to examine the front and back of the eye, aiding in the diagnosis of various conditions, and often involves scoring or grading for certain aspects like cell and flar

CONTACTS AND LOCATIONS:
Locations (1):
- Al Mustafa eye hospital lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No